CLINICAL TRIAL: NCT01009827
Title: Network-Wide Assessment of Current Health Status and Behavioral Risk Factors
Brief Title: Managerial Database II
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Other Study IDs: ATN 086
Record Dates: First submitted 2009-11-06; First posted 2009-11-09 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2016-03

CONDITIONS: HIV
Keywords: Medication adherence; Substance use; Sexual risk behaviors
MeSH Terms: conditions — Medication Adherence; Substance-Related Disorders | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- AMTU Clients: All HIV-infected adolescents and young adults engaged in care at the 15 sites and their affiliates who are between 12 and 24 years of age, inclusive, are aware of their HIV status and understand written and/or verbal English will be eligible for inclusion in the study. In addition, new patients who have their initial clinic visit within the enrollment period will also be eligible for participation.
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — Participants will have biomedical information extracted from their medical chart, will complete the ACASI questionnaire and have a face-to-face post-ACASI debriefing interview administered. Participants who do not have a documented HIV-1 viral load and/or CD4+ T-cells count from within the previous six months will also have venipuncture performed to obtain a blood sample for these tests to be performed.

SUMMARY:
This study will collect information on health status and risk behaviors, as well as basic demographic and biomedical information for a group of HIV positive adolescents receiving care at the ATN sites.

DETAILED DESCRIPTION:
The proposed study is a cross sectional study intended to be conducted at each of the 15 Adolescent Medicine Trials Units (AMTUs) participating in the ATN and to enroll all participating patients followed at each site. This approach will allow for the examination of the broad spectrum of youth participating in the ATN, including those newly entered into care.

Psychosocial and risk-taking behavioral data will be collected using Audio Compute-Assisted Self-Interview (ACASI); biomedical information will be collected through medical chart abstraction.

ELIGIBILITY:
Inclusion Criteria:

* Laboratory evidence of HIV-1 infection documented by a positive result on any of the following licensed tests at any time: Any HIV-1 antibody test confirmed by Western blot, HIV-1 culture, HIV-1 DNA PCR, or plasma HIV-1 RNA PCR > 1,000 copies/ml;
* Knowledge of HIV positive diagnoses;
* Age 12 years through 24 years, inclusive;
* Engaged in care at the AMTU or its affiliate and/or partnering clinic. Individuals will be considered to be engaged in care if:
* Diagnosed less than or equal to 12 months prior to the date of approval to generate the master list and has attended a minimum of one visit since diagnosis for the management of HIV disease or its sequelae; or
* Diagnosed more than 12 months prior to the date of approval to generate the master list and has had a minimum of one visit, as described above, within the past 12 months.
* Ability to understand written and/or verbal English
* Ability and willingness to provide signed consent/assent;
* Parental/legal guardian permission (if applicable)

Exclusion Criteria:

* Presence of serious psychiatric symptoms (e.g., active hallucinations, thought disorder) that would impair the individuals' ability to complete the study measures;
* Visibly distraught (e.g., suicidal, homicidal, exhibiting violent behavior); or
* Intoxicated or under the influence of alcohol or other substances at the time of consent/assent.

Ages: 12 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All HIV-infected adolescents and young adults engaged in care at the 15 sites and their affiliates who are between 12 and 24 years of age, inclusive, are aware of their HIV status and understand written and/or verbal English will be included in the master list from which the study sample will be derived.
Sampling Method: Non-Probability Sample
Enrollment: 1712 (Actual)
Dates: Start 2009-10; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Rates of adherence to medical regimens, sexual risk behavior, substance use and mental health concerns; basic demographic and biomedical data for adolescents and young adults with HIV infection engaged in care at the AMTUs. | within 2 weeks of enrollment

SECONDARY OUTCOMES:
To better understand the complex relationships between adherence to medical regimens, sexual risk behavior, substance use and mental health concerns, and basic demographic and biomedical data in adolescents and young adults with HIV infection. | 1.3 years

CONTACTS AND LOCATIONS:
Overall Officials: Heather Huszti, Ph.D., Study Chair — Adolescent Trials Network
Locations (15):
- United States (14):
  - Childrens Hospital Los Angeles, Los Angeles, California
  - University of California San Francisco, San Francisco, California
  - Childrens National Medical Center, Washington D.C., District of Columbia
  - Childrens Diagnostic & Treatment Center, Fort Lauderdale, Florida
  - University of Miami School of Medicine, Miami, Florida
  - University of South Florida, Tampa, Florida
  - Ruth M Rothstein CORE Center/ John H Stroger Jr Hospital, Chicago, Illinois
  - Childrens Memorial Hospital, Chicago, Illinois
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - University of Maryland, Baltimore, Maryland
  - Mount Sinai Medical Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Childrens Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Jude Childrens Research Hospital, Memphis, Tennessee
- University of Puerto Rico, San Juan, Puerto Rico

REFERENCES:
- See also: ATN Website — http://www.atnonline.org